CLINICAL TRIAL: NCT01315210
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of D-Ribose in Subjects With Fibromyalgia
Brief Title: D-Ribose for Fatigue in Subjects With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RiboCor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIOE 02C 010
Record Dates: First submitted 2011-03-10; First posted 2011-03-15 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Fatigue; D-Ribose
MeSH Terms: conditions — Fibromyalgia; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-Ribose (Experimental)
  Interventions: Drug: D-Ribose Powder
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Drug: D-Ribose Powder — 5 g TID for 12 Weeks
  Arms: D-Ribose
Dietary Supplement: Placebo Powder — 5 g TID for 12 Weeks
  Arms: Placebo

SUMMARY:
To evaluate the safety and to determine the efficacy of D-ribose for the amelioration of fatigue in subjects with fibromyalgia. This is a phase IIa, randomized, double-blind, placebo-controlled, multi-center, multiple dose study of D-ribose versus placebo administered at doses of 5 g three times a day (TID) over a 12-week period to subjects who are experiencing fatigue associated with a diagnosis of fibromyalgia.

ELIGIBILITY:
Major Inclusion Criteria:

* must have a diagnosis of primary fibromyalgia, as defined by the 1990 American College of Rheumatology (ACR) Criteria for the Classification of Fibromyalgia made at least 6 weeks prior to the Pretreatment Screening Visit;
* must have a score of ≥5 on the Subject's Assessment of Fatigue 11-point numerical rating scale (NRS) at the Pretreatment Screening and Baseline Visits;
* if taking acetaminophen or other non-opioid analgesics, NSAIDs, fibromyalgia medications, medications to induce sleep, or prednisone ≤ 10 mg (or equivalent dose of other glucocorticoids), must be on stable dose(s) for at least 4 weeks prior to the baseline visit;
* must have discontinued any ribose-containing products (including foods, drinks, and supplements) at least 4 weeks prior to the Pretreatment Baseline Visit.

Major Exclusion Criteria:

* current major depressive episode (MDE);
* has been diagnosed with any autoimmune disease;
* has been diagnosed with type I or type II diabetes;
* has a history of cancer, other than basal cell carcinoma, stage 1 squamous cell carcinoma or cervical carcinoma in situ, that has not been in remission for at least five years prior to the Pretreatment Screening Visit;
* has been diagnosed with chronic fatigue syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Subject's Assessment of Fatigue (NRS) | 12 Weeks

SECONDARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire | 12 Weeks
Multidimensional Fatigue Inventory | 12 Weeks
Subject's Global Impression of Change | 12 Weeks
SF-36 | 12 Weeks
Subject's Assessment of Pain Intensity (NRS) | 12 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Crofford, MD, Principal Investigator — University of Kentucky
Locations (9):
- United States (9):
  - Superior Research, LLC, Sacramento, California
  - Avail Clinical Research, DeLand, Florida
  - Renstar Medical Research, Ocala, Florida
  - University of Kentucky, Lexington, Kentucky
  - Columbia Medical Practice, Columbia, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Peters Medical Research, High Point, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania